CLINICAL TRIAL: NCT01520649
Title: A Phase 1B, Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose Escalation Study Evaluating the Safety, Tolerability, Pharmacokinetics (PK), and Pharmacodynamic (PD) Effect of NSI-189 Phosphate in Depression Patient Subjects
Brief Title: Multiple-Dose Pharmacokinetics (PK), and Pharmacodynamic (PD) Effect of NSI-189 Phosphate in Depression Patient Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neuralstem Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NS-2010-3
Record Dates: First submitted 2012-01-25; First posted 2012-01-30 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2012-11

CONDITIONS: Depression
Keywords: Neurogenesis; hippocampal stem cells; depression; stroke
MeSH Terms: conditions — Depression; Stroke | interventions — NSI-189; microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NSI-189 Phosphate (Experimental): There will be 3 ascending cohorts. The first cohort will be administered 40 mg once daily (q.d). The second cohort will be administered 40 mg twice daily (b.i.d). The third cohort will be administered 40 mg three times daily (t.i.d).
  Interventions: Drug: NSI-189 Phosphate
- microcrystalline cellulose capsules (Placebo Comparator): The first cohort will be administered 40 mg once daily (q.d). The second cohort will be administered 40 mg twice daily (b.i.d). The third cohort will be administered 40 mg three times daily (t.i.d).
  Interventions: Drug: microcrystalline cellulose capsules

INTERVENTIONS:
Drug: NSI-189 Phosphate — The first cohort will be administered 40 mg once daily (q.d). The second cohort will be administered 40 mg twice daily (b.i.d). The third cohort will be administered 40 mg three times daily (t.i.d).
  Arms: NSI-189 Phosphate
Drug: microcrystalline cellulose capsules — The first cohort will be administered 40 mg once daily (q.d). The second cohort will be administered 40 mg twice daily (b.i.d). The third cohort will be administered 40 mg three times daily (t.i.d).
  Arms: microcrystalline cellulose capsules

SUMMARY:
This is a Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose Escalation in depressed human subjects study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has the ability to understand the purpose and risks of the study and to provide signed and dated informed consent, authorizing to use of protected health information in accordance with national and local patient privacy regulations.
2. Males and females 18 to 60 years of age, inclusive, at the time of informed consent.
3. Diagnosis of major depressive disorder, recurrent, as per DSM-IV-TR criteria and confirmed by SCID-CT. Their major depressive episode must be confirmed via SCID mood module interview administered by remote, independent raters.

   Note: Both patients who are being treated with antidepressants and patients who are not on antidepressants but had a history of taking antidepressants are permitted in the study.
4. Montgomery-Asberg Depression Scale (MADRS) score of 15 to 30, inclusive, at Screening and baseline.
5. The following applies to female patients:Non-pregnant, non-lactating females of childbearing potential who agree to use medically acceptable forms of birth control (hormonal contraception, abstinence, diaphragm with spermicide, condom with spermicide, or intrauterine device) from Screening until the end-of-study.
6. The following applies to male subjects:

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2012-05; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Safety of drug assessed by number and severity of adverse events in drug vs placebo group | 28 days
  Values for vital signs, standard physical examination, ECG, EEG, standard clinical laboratory tests (hematology and biochemistry), standard neurological exam and the Columbia Suicide Severity Rating Scale will be compared between NSI 189 and placebo.

SECONDARY OUTCOMES:
Pharmacokinetics of NSI 189 will be determined by plasma sample collection at various timepoints pre, during and post dosing, measuring the concentration of drug over time. | 28 days
  Concentration of NSI 189 will be measured in plasma and standard pK values will be determined:AUC, Cmax, Tmax, T1/2, CL, Vz.

CONTACTS AND LOCATIONS:
Overall Officials: Karl Johe, PhD, Study Director — Neuralstem Inc.
Locations (1):
- California Clinical Trials, Glendale, California, United States

REFERENCES:
- [Background] Kessler RC, Berglund P, Demler O, Jin R, Koretz D, Merikangas KR, Rush AJ, Walters EE,Wang PS; National Comorbidity Survey Replication. The epidemiology of major depressive disorder: results from the National Comorbidity Survey Replication (NCS-R). JAMA. 2003 Jun 18;289(23):3095-105. PubMed PMID: 12813115. Deng W, Aimone JB, Gage FH. New neurons and new memories: how does adult hippocampal neurogenesis affect learning and memory? Nat Rev Neurosci. 2010 May;11(5):339-50. Epub 2010 Mar 31. Review. PubMed PMID: 20354534; PubMed Central PMCID: PMC2886712. DeCarolis NA, Eisch AJ. Hippocampal neurogenesis as a target for the treatment of mental illness: a critical evaluation. Neuropharmacology. 2010 May;58(6):884-93. Epub 2010 Jan 6. Review. PubMed PMID: 20060007; PubMed Central PMCID: PMC2839019. Marlatt MW, Lucassen PJ. Neurogenesis and Alzheimer's disease: Biology and pathophysiology in mice and men. Curr Alzheimer Res. 2010 Mar;7(2):113-25. Review.PubMed PMID: 19860727. Kernie SG, Parent JM. Forebrain neurogenesis after focal Ischemic and traumatic brain injury. Neurobiol Dis. 2010 Feb;37(2):267-74. Epub 2009 Nov 10. Review. PubMed PMID:19909815; PubMed Central PMCID: PMC2864918. Kempermann G, Krebs J, Fabel K. The contribution of failing adult hippocampalneurogenesis to psychiatric disorders. Curr Opin Psychiatry. 2008;21(3):290-5. PMID:18382230.